CLINICAL TRIAL: NCT04890249
Title: Clinical Investigation of the TECNIS® Intraocular Lens, Models C1V000 and C2V000
Brief Title: Clinical Investigation of Two Tecnis Investigational Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PCOL-102-AHSF
Record Dates: First submitted 2021-05-06; First posted 2021-05-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cataract; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational Lens Device #1 (Experimental): Investigational IOL Model C1V000
  Interventions: Device: Investigational IOL Model C1V000
- Investigational Lens Device #2 (Experimental): Investigational IOL Model C2V000
  Interventions: Device: Investigational IOL Model C2V000
- Control Lens (Active Comparator): Control IOL Model ICB00
  Interventions: Device: Control IOL Model ICB00

INTERVENTIONS:
Device: Investigational IOL Model C1V000 — IOL replaces the natural lens removed during cataract surgery.
  Arms: Investigational Lens Device #1
Device: Investigational IOL Model C2V000 — IOL replaces the natural lens removed during cataract surgery.
  Arms: Investigational Lens Device #2
Device: Control IOL Model ICB00 — IOL replaces the natural lens removed during cataract surgery.
  Arms: Control Lens

SUMMARY:
This study is a 6-month, prospective, multicenter, randomized (1:1:1), subject-masked and evaluator-masked, bilateral clinical investigation of the TECNIS IOL Models C1V000 and C2V000 versus the TECNIS Eyhance™ Model ICB00 IOL.

The study will be conducted at up to 15 sites in EU, AU, NZ and/or AP and will enroll up to 225 subjects to achieve approximately 67 bilaterally implanted subjects in each lens group. Allowing for 10% lost-to-follow-up, this will achieve approximately 60 evaluable subjects in each lens group at 1, 3, and 6 months. The eye implanted first will be considered the primary (monocular) study eye.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts or planned natural lens removal (due to immature cataract) for which phacoemulsification extraction and posterior IOL implantation have been planned for both eyes
* Cataractous lens changes, as demonstrated by best-corrected distance visual acuity (BCDVA) of 0.50 decimal or worse (6/12 or 20/40 Snellen) either with or without a glare source present (e.g., Brightness Acuity Tester) or with significant cataract-related visual symptoms in the opinion of the investigator
* Potential postoperative best-corrected distance visual acuity (BCDVA) of 0.66 decimal (6/9 or 20/30 Snellen) or better
* Corneal astigmatism:

  * Normal corneal topography
  * Predicted postoperative corneal astigmatism of less than 1.00 D in both eyes, including posterior corneal astigmatism (PCA)
* Clear intraocular media other than cataract
* Signed informed consent for participation in the study and data protection
* Availability, willingness, ability, and sufficient cognitive awareness to comply with examination procedures and study visits
* Ability to understand, read, and write English or the local language in which the informed consent and questionnaires are provided.

Exclusion Criteria:

* Requiring an intraocular lens power outside the available range of +14.0 D to +26.0 D
* Any clinically significant pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery, including prophylactic peripheral iridotomies and peripheral laser retinal repairs
* Corneal abnormalities such as stromal, epithelial, or endothelial dystrophies (e.g., any observed guttata) that are predicted to cause visual acuity losses to a level worse than 0.66 decimal (6/9 or 20/30 Snellen) during the study
* Irregular corneal astigmatism
* Inability to achieve keratometric stability for contact lens wearers
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level worse than 0.66 decimal (6/9 or 20/30 Snellen) during the study
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use during the course of the 6-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
* Poorly controlled diabetes
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.) Note: Controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable
* Known ocular disease or pathology that, in the opinion of the investigator,

  * may affect visual acuity
  * may require surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, uncontrolled glaucoma, etc.)
  * may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
* Pregnancy, planned pregnancy, presently lactating, or another condition associated with hormonal fluctuation that could lead to refractive changes
* Concurrent participation or participation within 60 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Monocular Photopic distance-corrected intermediate visual acuity | 6 months
Monocular Photopic best-corrected distance visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (8):
- Australia (7):
  - personalEYES Pty. Ltd., Burwood, New South Wales
  - Vision Eye Institute, Chatswood, New South Wales
  - George St Eye Centre, Sydney, New South Wales
  - Bondi Eye Doctors, Sydney, New South Wales
  - Newcastle Eye Hospital, Waratah, New South Wales
  - Sunshine Eye Clinic, Birtinya, Queensland
  - Queensland Eye Institute, South Brisbane, Queensland
- Auckland Eye Ltd, Remuera, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu